CLINICAL TRIAL: NCT06774391
Title: CARDIOVASCular Unexpected fiNdings in patiEnts Undergoing eXecution of PET/tc (CV-UNEXPET/TC)
Brief Title: CARDIOVASCular Unexpected fiNdings in patiEnts Undergoing eXecution of PET/tc
Acronym: CV-UNEXPET/TC
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CV-UNEXPET/TC
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-11

CONDITIONS: Cardiovascular Disease Other
Keywords: CIED; amyloidosis; cardiomyopathies; atrial fibrillation; PET/TC
MeSH Terms: conditions — Amyloidosis; Cardiomyopathies; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this single-center observational study is to retrospectively evaluate incidental findings at the cardiovascular level in a selection of patients referred to the O.U. of Nuclear Medicine of Policlinco S.Orsola-Malpighi who underwent a PET/CT investigation.

In particular, the present study is aimed to explore in such patients occasional findings of hypercapturing radiopharmaceutical findings specifically referred to:

* infection inflammatory processes of implantable cardiac devices (ICDs, pacemakers);
* phenomena affecting the atria during episodes of atrial fibrillation;
* infection and inflammatory processes of cardiovascular structures (endocarditis, myocarditis, pericarditis, amyloidosis).

Patients who performed PET/CT examination at the Sant'Orsola-Malpighi Nuclear Medicine O.U. during the period between 01/01/2017 and 31/12/2019 will be included in this registry. Any cardiovascular events that occurred within the Sant'Orsola-Malpighi Polyclinic setting and up to 3 months after the date of the PET/CT scan will be subsequently evaluated.

DETAILED DESCRIPTION:
The present study aims to investigate the role of PET/CT investigation in the detection of abnormal ancillary findings, in this case of the cardiovascular type. This aspect, at first glance of secondary importance with respect to the reasons why a patient undergoes this diagnostic examination, is actually of some importance, since early detection of some significant incidental findings (otherwise misrecognized because they are not related to any symptomatic cortex) can often negatively influence several patient-related factors:

* Response to therapy (e.g., chemotherapy);
* Comorbidities;
* Life expectancy;
* Quality of life.

All data of patients referred to the U.O. of Nuclear Medicine of Policlinico S.Orsola-Malpighi who underwent a PET/CT investigation from 01/01/2017 to 31/12/2019 will be collected. Of these patients, the biographical data, clinical news, biochemical tests, any other imaging investigations (CT, echocardiography, MRI) will be collected. Within the population, patients who, upon review and anonymization of PET/CT images, show significant radiotracer hyperfixation at the cardiovascular level will be identified. Incidental findings referable to:

* infection and inflammatory phenomena of implantable cardiac devices (ICDs, pacemakers);
* misdiagnosed episodes of atrial fibrillation;
* infection and phlogistic phenomena of cardiovascular structures (endocarditis, myocarditis, pericarditis, amyloidosis).

The computerized approach of the study involves the following steps. Starting from the computerized database that collects the main clinical-anamnestic information of all patients afferent to the Nuclear Medicine Cluster of Policlinico S.Orsola-Malpighi (ASTRIM), specific queries will be created for automatic filtering by keywords of only the patients of interest, specifically:

* For patients who carry intracardiac devices, selection will be by keywords such as "pacemaker," "defibrillators," "ICD"; "CIED."
* For patients with a history of amyloidosis or heart failure, selection is through keywords such as "amyloidosis" "heart failure."
* For patients with a history of atrial fibrillation, selection is through keywords such as "atrial fibrillation," "AF."

This initial search will be complemented by a second selection of patients whose PET/CT report contains keywords that may point to the presence of hypermetabolic findings at the cardiac level. By entering keywords such as "pacemaker," "device," "electrocatheter," "atrial," "atrial fibrillation," and "amyloidosis" on the ERIS computer system, it will be possible to quickly identify all patients with suspicious findings at the cardiac level and reported by the nuclear physician on the validated report. In addition, the names of patients with intracardiac devices followed up at the Cardio-Thoracic-Vascular Pole of Policlinico S.Orsola-Malpighi will be provided; of them, it will be possible to extrapolate those who underwent PET/CT during the period taken into consideration of the study. Therefore, it is estimated that from a total database of approximately 35,000-40,000 examinations, about a thousand patients will be selected through the procedures described above. From the excluded patients with sufficient recorded clinical data, control groups matched for age, sex, and indication for evaluation by PET/CT will be produced.

Therefore, an initial analysis will be conducted in describing the selected group of patients with cardiovascular-type findings, analyzing the uptake patterns and semi-quantitative parameters (Standardized Uptake Value, SUV) and comparing them with the control group.

Then we will conduct through computerized data from three company databases (ERIS, Online Medical Records and the Cardio-Thoracic-Vascular Pole Implantable Cardiac Device Carriers Registry), a maximum 3-month monitoring aimed at identifying any hospital admissions for cardiovascular reasons justified by the previously found PET/CT finding.

The following data will be evaluated for each patient:

* Current medical history/concurrent therapies
* Past concomitant therapies
* Laboratory tests
* Inclusion/exclusion criteria
* PET/CT examination. In the 3 months following the PET/CT investigation, any cardiovascular events occurring in that time window and recorded within the S.Orsola-Malpighi Polyclinic will be evaluated.

The study is observational, noninterventional in nature. Patients were treated according to clinical practice in accordance with the physician's judgment and the information in the Technical Data Sheet of each individual Radiopharmaceutical.

Descriptive analysis will be conducted using appropriate statistics: Student's t-test, chi-square test. Significance will be achieved with p-values<0.05. Data will be presented for the population considering all patients included in the study.

The objective of the study is to search for incidental findings in an unselected population of patients who have undergone a PET/CT investigation. The estimated sample size will be about 1,000 patients, drawn from a total database that should include the totality of PET/CT investigations performed at the O.U. of Nuclear Medicine in Bologna and is estimated at about 35,000-45,000 examinations.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to the U.O. of Nuclear Medicine of Policlinico S.Orsola-Malpighi who underwent a PET/CT investigation from 01/01/2017 to 31/12/2019.
* age > 18 years old

Exclusion Criteria:

* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who performed PET/CT examinations at the Sant'Orsola-Malpighi Nuclear Medicine OU in the period between 01/01/2017 and 31/12/2019. Based on the services provided, it is estimated about 35,000-45,000 total examinations. Of these, through the infortmatic approach described just above, only patients of interest will be selected: an estimated 1,000. It should be noted that in the event that each patient has performed more than one PET/CT scan for the purpose of the study, a different patient ID will be identified for each investigation performed.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of all incidental cardiovascular findings hypercapturing 18-fluorodeoxyglucose and not justified by history | At enrollment
  The primary objective of the study is to assess the prevalence of all incidental cardiovascular findings hypercapturing the radiopharmaceutical and not justified by history, with subsequent characterization of the sites in relation to the indication for performing PET-CT.

SECONDARY OUTCOMES:
incidence of hospitalization for cardiovascular causes in subjects with incidental findings hypercapturing the radiopharmaceutical, compared with subjects without such findings compared with negative subjects | From enrollment to 3 months after
  The secondary objective of the study is to evaluate the incidence of hospitalization for cardiovascular causes in subjects with incidental findings hypercapturing 18-FDG, compared with subjects without such findings compared with negative subjects. The analysis will be limited to patients followed at Policlinico S. Orsola Malpighi for a period of not less than 3 months after the PET/CT scan was performed, or who presented with a cardiovascular event within that time window.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Diemberger, Prof, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS - Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy